CLINICAL TRIAL: NCT03210441
Title: Evaluation of Eating Habits and Dysgeusia During Chemotherapy Treatment: a Prospective Cohort Study on Patients Affected by Breast Cancer
Brief Title: Evaluation of Eating Habits and Dysgeusia During Chemotherapy Treatment in Patients Affected by Breast Cancer
Acronym: CHANGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, LUCIA VASSALLI, MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP2488
Record Dates: First submitted 2017-06-15; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer; Dysgeusia; Eating Behavior; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Dysgeusia; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients affected by breast cancer and potentially treated with taxane chemotherapy
- Group 2: Patients affected by breast cancer and not potentially treated without taxane chemotherapy

SUMMARY:
In post-menopause women affected by breast cancer and treated with chemotherapy, overweight and obesity are considered both a risk factors as well as a negative prognostic factors since they increase the risk of early relapse and death. Furthermore, a decrease in weight may also occur during chemotherapy and is associated to a reduced quality of life and survival. Also, the majority of patients under chemotherapy refer dysgeusia, an alteration in taste that can determine food aversion, selection of hypercaloric food or reduced food introduction up to malnutrition. Our aim is to evaluate eating habits changes in patients affected by breast cancer and under chemotherapy treatment and to better understand how this alterations influence the quality of life, anxiety, depression and insomnia of patients as well as overall survival.

DETAILED DESCRIPTION:
INTRODUCTION

Overweight and obesity represent a risk factor for hormone dependent cancers such as breast, endometrium, ovarian, uterine and gastrointestinal cancer.

In particular, overweight and obesity are risk factors for breast cancer in post-menopause women since they are associated to higher level of circulating estrogens, insulin, insulin-like growth factor levels, leptin, adiponectin, growth factors (such as hepatocyte growth factor) and inflammatory cytokines (TNFα and Interleukin-6 (IL-6)). Moreover, they reduce sex hormone binding globulin (SHBG) plasma levels. Overweight and obesity are also negative prognostic factors for breast cancer in post-menopause women since they increase the risk of early relapse and death. An increased weight (2.5-6.2 Kg) is commonly reported during chemotherapy treatment in post-menopause women. This is due to increased appetite, hyperphagia and hydric retention associated with reduced metabolism and physic activities. However, the weight gain during therapy is still not recognised as a negative prognostic factor.

Furthermore, a decrease in weight may also occur during chemotherapy. This is mainly due to lower appetite and early satiety, dysgeusia, nausea and vomiting or intolerance to certain foods. Decreasing weight can determine less efficacy and tolerance in therapy, more complications/infections, more and longer hospitalisations and, as a consequence, a reduced quality of life and survival.

Dysgeusia is an alteration in taste that can determine food aversion, selection of hypercaloric food or reduced food introduction up to malnutrition. More than 75% of patients under chemotherapy refer dysgeusia; this is related to drugs (such as folic acid competitors, cyclophosphamide cisplatin and taxanes) and can last for weeks. ln particular, taxanes determine a peripheral nerves degeneration. The results are a metallic taste and an alteration in salted perception. In addition, they determine a dose-dependent chemotherapy-induced peripheral neuropathy (CIPN) with painful paraesthesia, total areflexia and muscular extremities weakness. Dysgeusia is an underestimated problem. Instrumental examinations and laboratory tests can be useful but they cannot replace a detailed medical history and a close physical examination associated with international validate questionnaires.

At the moment, no agreement was found on chemotherapy-induced dysgeusia prevention and therapy. Patients resolve this problems with cold food, candies before meals and sugary drinks and these behaviours lead to increasing in weight.

STUDY DESIGN

This is a prospective cohort study for the evaluation of eating habits changes and dysgeusia in patients with breast cancer during chemotherapy treatment. It will explore also the potential relations with anxiety, depression, insomnia and quality of life. These evaluations will be actuated using internationally validate questionnaires.

METHODS

This study is based on the collection of data with international validate questionnaires:

* Food frequency questionnaire (FFQ) and photography atlas
* Chemotherapy-induced taste alteration scale (CiTAS): evaluation of changes in taste.
* Functional assessment of cancer therapy (FACT_B): evaluation of quality of life for physical health, social and familiar health, emotional health, functional health and health in relation with the pathology.
* Beck depression inventory (BDI) and HADS: evaluation of depression presence and its intensity.
* Pittsburgh sleep quality index (PSQI) and insomnia severity index (ISI): evaluation of sleep quality.
* State and trait anxiety inventory (STAI-Y): evaluation of anxiety presence and its intensity.

STATISTICAL CONSIDERATIONS

Based on the proportion of the women in overweight before chemotherapy is 30% and the proportion of the women in overweight after chemotherapy is 50% (with a 5% α error and an 80% strength), the established number of patients to include in the study is 186. In prevision of a 10% loss of patients in follow-up, 204 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and post-menopause women with histologic diagnosis of invasive breast cancer surgically treated (all pT and all pN)
* Patients must provide written informed consent to be enrolled in the study

Exclusion Criteria:

* Locally extended or metastatic (M1) disease;
* Previous surgical or radio therapeutic treatment (up to one year before the selection) in oral or nasal region;
* Other serious medical conditions that can limit patient capability to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients affected by invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2014-05-06 (Actual); Primary Completion 2018-05-06 (Estimated); Study Completion 2018-05-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate eating habits changes in patients affected by breast cancer during chemotherapy treatment | From basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  Appearence of dysgeusia, asthenia, diarrhoea, decreased or increased appetite, mucositis, nausea, stypsis, vomiting and meteorism will be evaluated throught Food frequency questionaire (FFQ) compared to baseline (nefore chemotherapy)

SECONDARY OUTCOMES:
Evaluation of dysgeusia | From basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  Presence of changes in food taste (sweet, salt, bitter) and food smell compared to baseline in patients treated with taxanes throught the evaluation of a food questionnaire
Evaluation of weight alterations | From basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  Evaluation of the correlation between eating habits changes and dysgeusia with changes in weight through weight/height measurement and BMI calculation to evaluate the influence of eating habits changes and changes in weight on outcome in patients (relapse free interval (RFI) and overall survival (OS))
Evaluation of eating habits changes | from basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  Food frequency questionnaire (FFQ), chemotherapy-induced taste alteration scale questionnaire (CiTAS)
Evaluation of the impact of eating habits changes and dysgeusia on quality of life | from basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  functional assessment of cancer therapy questionnaire (FACT_B)
Evaluation of the impact of eating habits changes and dysgeusia on depression | from basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  beck depression inventory (BDI) and HADS test
Evaluation of the impact of eating habits changes and dysgeusia on insomnia | from basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  pittsburgh sleep quality index (PSQI) and insomnia severity index (ISI)
Evaluation of the impact of eating habits changes and dysgeusia on anxiety, depression | from basal visit and after every 3 months (during and post-chemotherapy) up to 12 months post- chemotherapy
  state and trait anxiety inventory (STAI-Y) will be administered to patients

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Vassalli, MD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinicrope FA, Dannenberg AJ. Obesity and breast cancer prognosis: weight of the evidence. J Clin Oncol. 2011 Jan 1;29(1):4-7. doi: 10.1200/JCO.2010.32.1752. Epub 2010 Nov 29. No abstract available. PMID 21115867
- [Background] Chlebowski RT, Aiello E, McTiernan A. Weight loss in breast cancer patient management. J Clin Oncol. 2002 Feb 15;20(4):1128-43. doi: 10.1200/JCO.2002.20.4.1128. PMID 11844838
- [Background] Goodwin PJ, Boyd NF. Body size and breast cancer prognosis: a critical review of the evidence. Breast Cancer Res Treat. 1990 Oct;16(3):205-14. doi: 10.1007/BF01806329. PMID 2085672
- [Background] Obermair A, Kurz C, Hanzal E, Bancher-Todesca D, Thoma M, Bodisch A, Kubista E, Kyral E, Kaider A, Sevelda P, et al. The influence of obesity on the disease-free survival in primary breast cancer. Anticancer Res. 1995 Sep-Oct;15(5B):2265-9. PMID 8572635
- [Background] Litton JK, Gonzalez-Angulo AM, Warneke CL, Buzdar AU, Kau SW, Bondy M, Mahabir S, Hortobagyi GN, Brewster AM. Relationship between obesity and pathologic response to neoadjuvant chemotherapy among women with operable breast cancer. J Clin Oncol. 2008 Sep 1;26(25):4072-7. doi: 10.1200/JCO.2007.14.4527. PMID 18757321
- [Background] Rosner GL, Hargis JB, Hollis DR, Budman DR, Weiss RB, Henderson IC, Schilsky RL. Relationship between toxicity and obesity in women receiving adjuvant chemotherapy for breast cancer: results from cancer and leukemia group B study 8541. J Clin Oncol. 1996 Nov;14(11):3000-8. doi: 10.1200/JCO.1996.14.11.3000. PMID 8918498
- [Background] Tredan O, Bajard A, Meunier A, Roux P, Fiorletta I, Gargi T, Bachelot T, Guastalla JP, Lallemand Y, Faure C, Perol D, Bachmann P. Body weight change in women receiving adjuvant chemotherapy for breast cancer: a French prospective study. Clin Nutr. 2010 Apr;29(2):187-91. doi: 10.1016/j.clnu.2009.08.003. Epub 2009 Aug 26. PMID 19713014
- [Background] Saquib N, Flatt SW, Natarajan L, Thomson CA, Bardwell WA, Caan B, Rock CL, Pierce JP. Weight gain and recovery of pre-cancer weight after breast cancer treatments: evidence from the women's healthy eating and living (WHEL) study. Breast Cancer Res Treat. 2007 Oct;105(2):177-86. doi: 10.1007/s10549-006-9442-2. Epub 2006 Nov 23. PMID 17123151
- [Background] Harvie MN, Campbell IT, Baildam A, Howell A. Energy balance in early breast cancer patients receiving adjuvant chemotherapy. Breast Cancer Res Treat. 2004 Feb;83(3):201-10. doi: 10.1023/B:BREA.0000014037.48744.fa. PMID 14758090
- [Background] Goodwin PJ, Ennis M, Pritchard KI, McCready D, Koo J, Sidlofsky S, Trudeau M, Hood N, Redwood S. Adjuvant treatment and onset of menopause predict weight gain after breast cancer diagnosis. J Clin Oncol. 1999 Jan;17(1):120-9. doi: 10.1200/JCO.1999.17.1.120. PMID 10458225
- [Background] Demark-Wahnefried W, Rimer BK, Winer EP. Weight gain in women diagnosed with breast cancer. J Am Diet Assoc. 1997 May;97(5):519-26, 529; quiz 527-8. doi: 10.1016/s0002-8223(97)00133-8. PMID 9145091
- [Background] Demark-Wahnefried W, Winer EP, Rimer BK. Why women gain weight with adjuvant chemotherapy for breast cancer. J Clin Oncol. 1993 Jul;11(7):1418-29. doi: 10.1200/JCO.1993.11.7.1418. PMID 8315439
- [Background] Demark-Wahnefried W, Hars V, Conaway MR, Havlin K, Rimer BK, McElveen G, Winer EP. Reduced rates of metabolism and decreased physical activity in breast cancer patients receiving adjuvant chemotherapy. Am J Clin Nutr. 1997 May;65(5):1495-501. doi: 10.1093/ajcn/65.5.1495. PMID 9129482
- [Background] Camoriano JK, Loprinzi CL, Ingle JN, Therneau TM, Krook JE, Veeder MH. Weight change in women treated with adjuvant therapy or observed following mastectomy for node-positive breast cancer. J Clin Oncol. 1990 Aug;8(8):1327-34. doi: 10.1200/JCO.1990.8.8.1327. PMID 2199619
- [Background] Chlebowski RT, Weiner JM, Reynolds R, Luce J, Bulcavage L, Bateman JR. Long-term survival following relapse after 5-FU but not CMF adjuvant breast cancer therapy. Breast Cancer Res Treat. 1986;7(1):23-30. doi: 10.1007/BF01886732. PMID 3516262
- [Background] Hoskin PJ, Ashley S, Yarnold JR. Weight gain after primary surgery for breast cancer--effect of tamoxifen. Breast Cancer Res Treat. 1992;22(2):129-32. doi: 10.1007/BF01833342. PMID 1391977
- [Background] Fisher B, Dignam J, Bryant J, DeCillis A, Wickerham DL, Wolmark N, Costantino J, Redmond C, Fisher ER, Bowman DM, Deschenes L, Dimitrov NV, Margolese RG, Robidoux A, Shibata H, Terz J, Paterson AH, Feldman MI, Farrar W, Evans J, Lickley HL. Five versus more than five years of tamoxifen therapy for breast cancer patients with negative lymph nodes and estrogen receptor-positive tumors. J Natl Cancer Inst. 1996 Nov 6;88(21):1529-42. doi: 10.1093/jnci/88.21.1529. PMID 8901851
- [Background] Day R, Ganz PA, Costantino JP, Cronin WM, Wickerham DL, Fisher B. Health-related quality of life and tamoxifen in breast cancer prevention: a report from the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Clin Oncol. 1999 Sep;17(9):2659-69. doi: 10.1200/JCO.1999.17.9.2659. PMID 10561339
- [Background] Powles T, Eeles R, Ashley S, Easton D, Chang J, Dowsett M, Tidy A, Viggers J, Davey J. Interim analysis of the incidence of breast cancer in the Royal Marsden Hospital tamoxifen randomised chemoprevention trial. Lancet. 1998 Jul 11;352(9122):98-101. doi: 10.1016/S0140-6736(98)85012-5. PMID 9672274
- [Background] Baum M, Buzdar A, Cuzick J, Forbes J, Houghton J, Howell A, Sahmoud T; ATAC (Arimidex, Tamoxifen Alone or in Combination) Trialists' Group. Anastrozole alone or in combination with tamoxifen versus tamoxifen alone for adjuvant treatment of postmenopausal women with early-stage breast cancer: results of the ATAC (Arimidex, Tamoxifen Alone or in Combination) trial efficacy and safety update analyses. Cancer. 2003 Nov 1;98(9):1802-10. doi: 10.1002/cncr.11745. PMID 14584060
- [Background] Francini G, Petrioli R, Montagnani A, Cadirni A, Campagna S, Francini E, Gonnelli S. Exemestane after tamoxifen as adjuvant hormonal therapy in postmenopausal women with breast cancer: effects on body composition and lipids. Br J Cancer. 2006 Jul 17;95(2):153-8. doi: 10.1038/sj.bjc.6603258. PMID 16835585
- [Background] Sestak I, Harvie M, Howell A, Forbes JF, Dowsett M, Cuzick J. Weight change associated with anastrozole and tamoxifen treatment in postmenopausal women with or at high risk of developing breast cancer. Breast Cancer Res Treat. 2012 Jul;134(2):727-34. doi: 10.1007/s10549-012-2085-6. Epub 2012 May 16. PMID 22588672
- [Background] Blackburn GL, Wang KA. Dietary fat reduction and breast cancer outcome: results from the Women's Intervention Nutrition Study (WINS). Am J Clin Nutr. 2007 Sep;86(3):s878-81. doi: 10.1093/ajcn/86.3.878S. PMID 18265482
- [Background] Hovan AJ, Williams PM, Stevenson-Moore P, Wahlin YB, Ohrn KE, Elting LS, Spijkervet FK, Brennan MT; Dysgeusia Section, Oral Care Study Group, Multinational Association of Supportive Care in Cancer (MASCC)/International Society of Oral Oncology (ISOO). A systematic review of dysgeusia induced by cancer therapies. Support Care Cancer. 2010 Aug;18(8):1081-7. doi: 10.1007/s00520-010-0902-1. Epub 2010 May 22. PMID 20495984
- [Background] Ravasco P. Aspects of taste and compliance in patients with cancer. Eur J Oncol Nurs. 2005;9 Suppl 2:S84-91. doi: 10.1016/j.ejon.2005.09.003. PMID 16437761
- [Background] Bernhardson BM, Tishelman C, Rutqvist LE. Self-reported taste and smell changes during cancer chemotherapy. Support Care Cancer. 2008 Mar;16(3):275-83. doi: 10.1007/s00520-007-0319-7. Epub 2007 Aug 21. PMID 17710445
- [Background] Hong JH, Omur-Ozbek P, Stanek BT, Dietrich AM, Duncan SE, Lee YW, Lesser G. Taste and odor abnormalities in cancer patients. J Support Oncol. 2009 Mar-Apr;7(2):58-65. PMID 19408458
- [Background] Gamper EM, Giesinger JM, Oberguggenberger A, Kemmler G, Wintner LM, Gattringer K, Sperner-Unterweger B, Holzner B, Zabernigg A. Taste alterations in breast and gynaecological cancer patients receiving chemotherapy: prevalence, course of severity, and quality of life correlates. Acta Oncol. 2012 Apr;51(4):490-6. doi: 10.3109/0284186X.2011.633554. Epub 2011 Nov 30. PMID 22129358
- [Background] Augusto C, Pietro M, Cinzia M, Sergio C, Sara C, Luca G, Scaioli V. Peripheral neuropathy due to paclitaxel: study of the temporal relationships between the therapeutic schedule and the clinical quantitative score (QST) and comparison with neurophysiological findings. J Neurooncol. 2008 Jan;86(1):89-99. doi: 10.1007/s11060-007-9438-8. Epub 2007 Jul 5. PMID 17611715
- [Background] Lee JJ, Swain SM. Peripheral neuropathy induced by microtubule-stabilizing agents. J Clin Oncol. 2006 Apr 1;24(10):1633-42. doi: 10.1200/JCO.2005.04.0543. PMID 16575015
- [Background] Heckmann JG, Heckmann SM, Lang CJ, Hummel T. Neurological aspects of taste disorders. Arch Neurol. 2003 May;60(5):667-71. doi: 10.1001/archneur.60.5.667. No abstract available. PMID 12756129
- [Background] Cella D, Peterman A, Hudgens S, Webster K, Socinski MA. Measuring the side effects of taxane therapy in oncology: the functional assesment of cancer therapy-taxane (FACT-taxane). Cancer. 2003 Aug 15;98(4):822-31. doi: 10.1002/cncr.11578. PMID 12910528
- [Background] Kano T, Kanda K. Development and validation of a chemotherapy-induced taste alteration scale. Oncol Nurs Forum. 2013 Mar;40(2):E79-85. doi: 10.1188/13.ONF.E79-E85. PMID 23448748
- [Background] Strasser F, Demmer R, Bohme C, Schmitz SF, Thuerlimann B, Cerny T, Gillessen S. Prevention of docetaxel- or paclitaxel-associated taste alterations in cancer patients with oral glutamine: a randomized, placebo-controlled, double-blind study. Oncologist. 2008 Mar;13(3):337-46. doi: 10.1634/theoncologist.2007-0217. PMID 18378545
- [Background] Rehwaldt M, Wickham R, Purl S, Tariman J, Blendowski C, Shott S, Lappe M. Self-care strategies to cope with taste changes after chemotherapy. Oncol Nurs Forum. 2009 Mar;36(2):E47-56. doi: 10.1188/09.onf.e47-e56. PMID 19273394
- [Background] Speck RM, DeMichele A, Farrar JT, Hennessy S, Mao JJ, Stineman MG, Barg FK. Taste alteration in breast cancer patients treated with taxane chemotherapy: experience, effect, and coping strategies. Support Care Cancer. 2013 Feb;21(2):549-55. doi: 10.1007/s00520-012-1551-3. Epub 2012 Aug 5. PMID 22864536
- [Background] Buttigliero C, Monagheddu C, Petroni P, Saini A, Dogliotti L, Ciccone G, Berruti A. Prognostic role of vitamin d status and efficacy of vitamin D supplementation in cancer patients: a systematic review. Oncologist. 2011;16(9):1215-27. doi: 10.1634/theoncologist.2011-0098. Epub 2011 Aug 11. PMID 21835895
- [Result] Ewertz M, Jensen MB, Gunnarsdottir KA, Hojris I, Jakobsen EH, Nielsen D, Stenbygaard LE, Tange UB, Cold S. Effect of obesity on prognosis after early-stage breast cancer. J Clin Oncol. 2011 Jan 1;29(1):25-31. doi: 10.1200/JCO.2010.29.7614. Epub 2010 Nov 29. PMID 21115856